CLINICAL TRIAL: NCT03938779
Title: Pelvic Floor Muscle Training and Stress Urinary Incontinence in Elite Athletes . Clinical Trial
Brief Title: Stress Urinary Incontinence in Elite Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Telma Pires, principal investigator, University of Trás-os-Montes and Alto Douro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 25/2017
Record Dates: First submitted 2019-04-25; First posted 2019-05-06 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Floor Disorders
Keywords: Elite Athletes; Volleyball; Pelvic Floor Muscle Training
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Volleyball team will be evaluated in two moments, at the beginning and 4 months after the PFMT. After 4 months, to compare with the control group and to evaluate if there are differences between groups, namely muscle strength
Who Masked: Participant
Masking Description: The participants do not know that there is a control group and an intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pelvic Floor Muscle Training (PFMT) (Experimental): Experimental group will perform for 4 months a PFMT
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT)
- Pad test (Experimental): The experimental and control group will perform the pad test twice. At the beginning of the evaluation and 4 months after the PFMT. The modified pad test, has the durability of a workout (2h30min)
  Interventions: Diagnostic Test: Pad test
- Kings Health Questionnaire (No Intervention): Kings Health Questionnaire to assess the impact of urinary incontinence on quality of life of women. Both groups will complete the questionnaire.
- perineometer (No Intervention): Both groups will perform perineometry at baseline and 4 months after

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training (PFMT) — PFMT is a protocol of exercises for prevention and treatment for Stress Urinary Incontinence in elite females athletes, volleyball team
  Arms: Pelvic Floor Muscle Training (PFMT)
Diagnostic Test: Pad test — Pad test is a standardised test for quantifying urine loss. Pad test is not invasive and provide an easy, inexpensive and objective assessment of urine loss.
  Arms: Pad test

SUMMARY:
A protocol of pelvic floor muscles training (PFMT) in elite athletes was applied. They will do it for 4 months. Then re-evaluated.

DETAILED DESCRIPTION:
The athletes of the Portuguese national female's volleyball team were evaluated through perineometry, pad-test and Kings health questionnaire. They were taught a plan of pelvic floor muscles training (PFMT) to perform for 4 months. After this time they will be re-evaluated with the same measuring instruments.

ELIGIBILITY:
Inclusion Criteria:

* Elite female athletes
* Nulliparous
* Volleyball team.

Exclusion Criteria:

* Inability to contract the PFM, elderly
* Prolapse of the pelvic organs.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women have a predisposition to stress urinary incontinence, caused by high-impact exercises
Enrollment: 15 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-08-04 (Estimated)

PRIMARY OUTCOMES:
Pad-test (Short-term) | 2 hour 30 min
  The pad test is a standardised test for quantifying urine loss.

OTHER OUTCOMES:
Kings Health Questionnaire (KHQ) | 10 minutes
  Was constructed in order to assess the impact of urinary incontinence on quality of life women, also evaluating urinary symptoms and subjective measures of severity. The KHQ is composed of 21 items investigating nine domains and it evaluates the agreement of the subjects on a 4- and 5- option Likert scale: general health perceptions (1item), incontinence impact (1 item), role limitations (2 items), physical limitations (2 items), social limitations (2 items), personal relationships (3 items), emotions (3 items), sleep and energy (2 items) and severity measures (5 items). Additionally, it has an independent subscale designed as a Symptom Severity Scale, which contains 11 items, measuring the presence and severity of urinary symptoms (Appendix 5). The KHQ scored from a minimum of 0 (best QoL) to a maximum of 100 (worst QoL), scored by every domain and by their global score. Scores of independent subscale (Symptom Severity Scale) was calculated in the same way.

CONTACTS AND LOCATIONS:
Locations (1):
- Telma Filipa Rodrigues Pereira Pires, Vila Real, Trás-os-Montes E Alto Douro, Portugal

IPD SHARING:
Plan to Share IPD: No
Urinary incontinence is a public health problem, which we must combat intervention measures and publication of clinical trials to prevent and treat urinary incontinence. The PFMT is the first line treatment advised by recent literature.

REFERENCES:
- [Result] Oliveira M, Ferreira M, Azevedo MJ, Firmino-Machado J, Santos PC. Pelvic floor muscle training protocol for stress urinary incontinence in women: A systematic review. Rev Assoc Med Bras (1992). 2017 Jul;63(7):642-650. doi: 10.1590/1806-9282.63.07.642. PMID 28977091
- [Result] Morkved S, Bo K. Effect of pelvic floor muscle training during pregnancy and after childbirth on prevention and treatment of urinary incontinence: a systematic review. Br J Sports Med. 2014 Feb;48(4):299-310. doi: 10.1136/bjsports-2012-091758. Epub 2013 Jan 30. PMID 23365417
- [Result] Da Roza T, de Araujo MP, Viana R, Viana S, Jorge RN, Bo K, Mascarenhas T. Pelvic floor muscle training to improve urinary incontinence in young, nulliparous sport students: a pilot study. Int Urogynecol J. 2012 Aug;23(8):1069-73. doi: 10.1007/s00192-012-1759-2. Epub 2012 May 3. PMID 22552685